

## TRIAL STATISTICAL ANALYSIS PLAN

c44703258-02

BI Trial No.: 1346-0011 Title: A phase III randomized, double-blind, placebo-controlled, parallel group trial to examine the efficacy and safety of iclepertin once daily over 26 week treatment period in patients with schizophrenia (CONNEX-1) **Investigational** Iclepertin **Product(s):** Responsible trial statistician(s): Phone: Fax: **Date of statistical** 25 Oct 2024 analysis plan: Version: 2 **** Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights

reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

001-MCS-50-415\_RD-01 (3.0) / Saved on: 18 Jan 2021

| 1. | TABLE OF CONTENTS |
|----------------|--------------------------------------------------|
| TITLE PA | GE1 |
| 1. | TABLE OF CONTENTS2 |
| LIST OF T | ΓABLES AND FIGURES4 |
| 2. | LIST OF ABBREVIATIONS5 |
| 3. | INTRODUCTION7 |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY8 |
| 5. | ENDPOINTS(S)9 |
| 5.1 | PRIMARY ENDPOINT(S)9 |
| <b>5.2</b> | SECONDARY ENDPOINT(S)9 |
| 5.2.1 | Key secondary endpoint(s)9 |
| 5.2.2 | Secondary endpoint(s)9 |
| 6. | GENERAL ANALYSIS DEFINITIONS |
| 6.1 | TREATMENT(S)14 |
| <b>6.2</b> | IMPORTANT PROTOCOL DEVIATIONS14 |
| 6.3 | INTERCURRENT EVENTS |
| 6.4 | SUBJECT SETS ANALYSED18 |
| | HANDI ING OF MICCING DATA AND OUT IEDG |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS |
| 6.7 | BASELINE, TIME WINDOWS AND CALCULATED VISITS21 |
| <b>7.</b> | PLANNED ANALYSIS |
| 7.1 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS25 |
| 7.2 | CONCOMITANT DISEASES AND MEDICATION25 |
| 7.3 | TREATMENT COMPLIANCE |
| 7.4<br>7.4.1 | PRIMARY ENDPOINT ANALYSIS |
| 7.4.1 | Primary analysis20 |
| 7.5 | SECONDARY ENDPOINT ANALYSIS |
| 7.5.1 | Key secondary endpoint analysis |
| 7.5.1.1 | Primary analysis |
| 752 | (Other) Secondary and reint analysis |
| 7.5.2 | (Other) Secondary endpoint analysis |
| 7.7 | EXTENT OF EXPOSURE33 |
| <b>7.7 7.8</b> | SAFETY ANALYSIS 33 |
| 7.8.1 | Adverse events 33 |
| 7.8.2 | Laboratory data 40 |

Boehringer Ingelheim TSAP for BI Trial No: 1346.11

**** c44703258-02

| 1 , | | • |
|------------|-----------------------------------------------|----|
| 7.8.3 | Vital signs | 40 |
| 7.8.4 | ECG | |
| <b>7.9</b> | OTHER ANALYSES | |
| 8. | TIMEPOINT OF RELEASE OF TREATMENT INFORMATION | 42 |
| 9. | REFERENCES | 43 |
| 11. | HISTORY TABLE | 55 |
| 11. | HIGIORI TADLE | 33 |

Table 11: 1

Proprietary confidential information © 2024 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# LIST OF TABLES AND FIGURES

| Table 6.1: 1 | Treatment descriptions |
|---|---|
| Table 6.1: 2 | Analysing treatment periods (same for all treatment groups)14 |
| Table 6.3: 1 | Definition and technical specification of intercurrent events15 |
| Figure 6.3: 1 | On-/off-treatment status of the study medication for efficacy analysis after |
| | ICEs |
| Table 6.6: 1 | PRECIS minimum non-missing items required for total/domain score |
| | calculation21 |
| Table 6.7: 1 | Analysis visit windows for MCCB, VRFCAT, SCoRS, and PANSS22 |
| Table 6.7: 2 | Analysis visit windows for PRECIS, EQ-5D-5L (patient)22 |
| Table 6.7: 3 | Analysis visit windows for Tower of London, SDS, EQ-5D-5L (caregiver), |
| | SPGI-S, SCQ |
| Table 6.7: 4 | Analysis visit windows for CGI-S |
| Table 6.7: 5 | Analysis visit windows for PGI-S |
| Table 6.7: 6 | Analysis visit windows for SAS/BARS/AIMS23 |
| Table 6.7: 7 | Analysis visit windows for clinical laboratory evaluations (on-treatment |
| | period)23 |
| Table 6.7: 8 | Analysis visit windows for weight and vital signs (on-treatment period)23 |
| Table 6.7: 9 | Analysis visit windows for Ophthalmological variables24 |
| Table 7.8.1: 1 | MedDRA preferred terms for user-defined AE categories of AEs suggestive |
| | of abuse potential or related to CNS depressant effects |
| Table 7.8.1: 2 | MedDRA preferred terms for BIcMQ of Decreased haemoglobin and |
| | anaemia (incl. non-haematological causes) |
| Table 7.8.1: 3 | MedDRA preferred terms for user-defined AE category of Drowsiness38 |
| Table 7.8.1: 4 | MedDRA preferred terms for user-defined AE categories of sleep disorder |
| | AEs |

History table ......55

# 2. LIST OF ABBREVIATIONS

| Term | Definition / description |
|---|---|
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| AIMS | Abnormal Involuntary Movement Scale |
| ANCOVA | Analysis of Covariance |
| BARS | Barns Akathisia Rating Scale |
| CGI-C | Clinical Global Impression of Change |
| CGI-S | Clinical Global Impression of Severity |
| CIAS | Cognitive Impairment Associated with Schizophrenia |
| C-SSRS | Columbia Suicidality Severity Rating Scale |
| CTP | Clinical Trial Protocol |
| EQ-5D VAS | EQ-5D Visual Analogue Scale |
| EQ-5D-5L | EuroQol-5-Dimension-5-Level |
| HCRU | Health Care Resource Utilization |
| ICE | Intercurrent Event |
| iPD | Important Protocol Deviation |
| J2R | Jump to Reference |
| MATRICS | Measurement and Treatment Research to Improve Cognition in Schizophrenia |
| MCCB | MATRICS Consensus Cognitive Battery |
| MedDRA | Medical Dictionary for Drug Regulatory Activities |
| MI | Multiple Imputation |
| MMRM | Mixed-effects Model for Repeated Measures |
| PANSS | Positive and Negative Syndrome Scale |
| PGI-C | Patient Global Impression of Change |
| PGI-S | Patient Global Impression of Severity |
| PK | Pharmacokinetics |
| PRECIS | Patient Reported Experience of Cognitive Impairment in Schizophrenia |
| REML | Restricted Maximum Likelihood |
| REP | Residual Effect Period |
| SAS | Simpson Angus Scale |

| Term | Definition / description |
|--------|-----------------------------------------------------|
| SCoRS | Schizophrenia Cognition Rating Scale |
| SCQ | Schizophrenia Caregiver Questionnaire |
| SDS | Sheehan Disability Score |
| SPGI-C | Study Partner Impression of Change |
| SPGI-S | Study Partner Global Impression of Severity |
| ToL | Tower of London |
| VRFCAT | Virtual Reality Functional Capacity Assessment Tool |

#### 3. INTRODUCTION

As per International Conference on Harmonisation (ICH) E9, the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This Trial Statistical Analysis Plan (TSAP) assumes familiarity with the Clinical Trial Protocol (CTP), including Protocol Amendments. In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomization.

SAS® Version 9.4 will be used for all analyses if not otherwise specified. Pheonix WinNonlin<sup>TM</sup> Version 8.1 will be used for pharmacokinetic (PK) analyses.

## 4. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

For the further endpoint of change from screening Visit 1a in PRECIS individual items and domain scores at Week 24, only the PRECIS domain scores will be analyzed, and the PRECIS individual items will not be analyzed.

Definition of baseline for the assessments of efficacy, PANSS and C-SSRS will include assessments up to but no later than the day of the first administration of study medication.

## 5. ENDPOINTS(S)

## 5.1 PRIMARY ENDPOINT(S)

The primary endpoint is

• Change from baseline in MCCB overall composite T-score at Week 26.

MCCB assessments are planned to be performed at screening (Visit 1), baseline (Visit 2), Week 12 (Visit 6), and Week 26 (Visit 11/EOT) or any early end of treatment visit.

Any post-baseline MCCB assessments performed within 28 days of the previous assessment will be considered invalid because of potential practice effects and will be excluded prior to any subsequent data handling and therefore from the planned analyses (5).

The MCCB overall composite T-score will be derived from seven domain scores from a total of ten tests (see CTP Table 5.1: 1). A larger MCCB overall composite T-score indicates better cognition.

## 5.2 SECONDARY ENDPOINT(S)

## 5.2.1 Key secondary endpoint(s)

The key secondary endpoints are:

- Change from baseline in Schizophrenia Cognitive Rating Scale (SCoRS) interviewer total score at Week 26
- Change from baseline in Virtual Reality Functional Capacity Assessment Tool (VRFCAT) adjusted total time T-score at Week 26.

A lower rating in SCoRS reflects a lesser degree of impairment. A higher T-score in VRFCAT indicates a better functional outcome.

The endpoints will be used as defined in CTP Section 5.

## 5.2.2 Secondary endpoint(s)

The other secondary endpoints are:

- Change from baseline in the T-score of the number of correct responses on Tower of London (ToL) at Week 26
- Change from screening Visit 1a in Patient Reported Experience of Cognitive Impairment in Schizophrenia (PRECIS) total score at Week 24

A higher T-score in ToL indicates a better outcome. A lower score in PRECIS corresponds to a better patient experience.

The endpoints will be used as defined in CTP Section 5.







#### 6. GENERAL ANALYSIS DEFINITIONS

### 6.1 TREATMENT(S)

For basic study information on treatments to be administered, assignment of treatment groups, select of doses, see CTP Section 4.

Table 6.1: 1 lists the two treatment groups in this study. Table 6.1: 2 defines the analysing treatment period for safety analyses. For this study, the residual effect period (REP) is defined as 12 days after the last dose of trial medication.

Table 6.1: 1 Treatment descriptions

| Long Name | Short Name |
|---------------------|------------------|
| Placebo | Placebo |
| Iclepertin 10 mg QD | Iclepertin 10 mg |

Table 6.1: 2 Analysing treatment periods (same for all treatment groups)

| Analysing Treatment<br>Period | Start Date | End Date |
|---|---|---|
| Screening period | Date of informed consent | Date of the first treatment administration – 1 day |
| On-treatment period | Date of the first treatment administration | Date of the last treatment administration + REP |
| Post-treatment period | Date of the last treatment administration + REP + 1 day | Date of the last per protocol visit |

REP is the residual effect period which is defined as 12 days after the last dose of trial treatment.

## 6.2 IMPORTANT PROTOCOL DEVIATIONS

Handling of iPDs in analyses is described in the iPD specification document and stored in the Trial Master File (TMF) in the electronic Document Management System (eDMS).

#### 6.3 INTERCURRENT EVENTS

Definition and technical specification of protocol defined intercurrent events (ICEs) are listed in <u>Table 6.3: 1</u>. In general, when handled under the hypothetical approach, data collected during the off-treatment period of an ICE will be considered irrelevant to the estimand and excluded from the analysis. While off-treatment data will be excluded, the patient will still be considered as on-treatment (hypothetically) from an analysis perspective by the statistical models, and during any imputations.

For an ICE of temporary treatment discontinuation or interruptions, the off-treatment period spans from the last treatment administration prior to the interruption + REP to the restart of

the study medication. For an ICE of early permanent treatment discontinuation, the off-treatment period starts from the last treatment administration + REP. <u>Figure 6.3: 1</u> illustrates the on-/off-treatment status after each type of ICEs. When there is more than one ICE of early permanent treatment discontinuation, any treatment policy ICE take precedence in data and analysis handling over any hypothetical ICE.

ICEs of change in concomitant therapies and other ICEs will always be considered as part of the treatment policy in the primary and all supplementary estimands. ICEs of this category will not affect the on-/off- treatment status which is only determined by changes in the study medication. These ICEs will be listed and summarized descriptively but will not be explicitly accounted for in the inferential analysis of efficacy.

Table 6.3: 1 Definition and technical specification of intercurrent events

| Type of<br>Intercurrent<br>Event | Definition and Documentary<br>Sources | Handling under the<br>Primary Estimand |
|---|---|---|
| Temporary Tr | eatment Discontinuations or Interruption | ons |
| Exacerbation or acute episode of schizophrenia resulting in interruption of treatment | Identified from data collected in the Temporary Trial Treatment Discontinuation and Adverse Event pages of the CRF: - Temporary discontinuation of trial treatment reported with reason being "Adverse Event", and - AE category reported as "Schizophrenia Relapse" or MedDRA preferred term coded as "Schizophrenia" | Treatment policy |
| Temporary<br>treatment<br>discontinuation or<br>interruption due to<br>other reasons | Identified from data collected in the Temporary Discontinuation page of the CRF. | Hypothetical – only data collected from the end of REP after the interruption, to end of the interruption will be subject to exclusion from the analysis |
| Temporary<br>treatment-switch<br>due to dispensation<br>error | Identified from the dispensation records. Temporary treatment-switch will be handled as temporary interruptions in the same way for both directions (iclepertin to placebo or placebo to iclepertin) | Hypothetical – only data collected from the end of REP after the treatment switch, to end of the treatment switch will be subject to exclusion from the analysis |
| Early Permanent Treatment Discontinuation | | |

| Exacerbation or | Identified from data collected in the | Treatment policy |
|---|---|---|
| acute episode of | Adverse Event page of the CRF: | Treatment poncy |
| schizophrenia<br>resulting in early<br>termination of<br>treatment | - "Drug Withdrawn" reported in<br>the Action Taken with Study<br>Treatment field, and | |
| | - Category reported as "Schizophrenia Relapse" or MedDRA preferred term coded as "Schizophrenia" | |
| Investigator assessed drug- | Identified from data collected in the Adverse Event page of the CRF: | Treatment policy |
| related adverse<br>events which lead<br>to early termination<br>of study | - "Drug Withdrawn" reported in<br>the Action Taken with Study<br>Treatment field, and | |
| medication | - "Yes" reported in the<br>Relationship to Study Treatment<br>field | |
| Protocol-defined<br>drug withdrawal<br>due to treatment –<br>haemoglobin<br>decrease | Identified from data collected in the End of Treatment and Adverse Event pages of the CRF and laboratory data: - Subject who did not complete the planned treatment period as reported in the End of Treatment page with reason being "Adverse Event", and - AE indicating haemoglobin decrease with action taken being "Drug Withdrawn" | Treatment policy |
| Protocol-defined drug withdrawal due to treatment – CYP3A4 inhibitors or CYP3A4 sensitive drugs with NTI | Identified from data collected in the End of Treatment page of the CRF: - Subject who did not complete the planned treatment period as reported in the End of Treatment page with "Protocol Deviation" as the reason, and - Use of CYP3A4 inhibitors or CYP3A4 sensitive drugs with NTI specified as the detailed reason of discontinuation | Treatment policy |
| Early termination of study | Identified from data collected in the End of Treatment page of the CRF: | Hypothetical |

| medication due to other AEs | - Subject who did not complete the planned treatment period as reported in the End of Treatment page with reason being "Adverse Event" and not otherwise covered by any of the ICEs above. | |
|---|---|---|
| Early termination of study medication due to perceived lack of efficacy | Identified from data collected in the End of Treatment page of the CRF: - Subject who did not complete the planned treatment period as reported in the End of Treatment page with reason being "Perceived Lack of Efficacy". | Hypothetical |
| Early termination of study medication due to other reasons | Identified from data collected in the End of Treatment page of the CRF: - Subject who did not complete the planned treatment period as reported in the End of Treatment page for reasons not covered by any of the ICEs above. | Hypothetical |
| Change in Co. | ncomitant Therapies and Other ICEs | |
| Change in background medication | Identified from data collected in the Concomitant Medications page of the CRF: - Start of a new or stop of an ongoing antipsychotic, benzodiazepines (or derivatives), anticholinergics, antiepileptics, or antidepressants during the ontreatment period, or - Change of dosage or dosing | Treatment policy |
| | frequencies of an on-going antipsychotic, benzodiazepines (or derivatives), anticholinergics, antiepileptics, or antidepressants during the on-treatment period See <u>Table 10.7: 1</u> for definitions of antipsychotics, benzodiazepines (or derivatives), anticholinergics, antiepileptics, and antidepressants. | |
| Change in psychotherapy | Identified from data collected in the Psychotherapy page of the CRF: | Treatment policy |

| | - Change in frequency, setting or session of a psychotherapy during the on-treatment period | |
|---|---|---|
| Change in other non-pharmacological therapy | Identified from data collected in the Concomitant Non-Drug Therapies page of the CRF: - Start of a new non-drug therapy or stop of an on-going non-drug therapy during the on-treatment period | Treatment policy |
| Change in study partner in the assessment of functional capacity, e.g. SCoRS | Identified from data collected in the Study Partner Informed Consent page of the CRF and date/time of SCoRS assessments: - Any new study partner informed consent signed between the baseline SCoRS assessment and the SCoRS assessment being considered | Treatment policy – relevant only to endpoints from the SCoRS assessment |

Figure 6.3: 1 On-/off-treatment status of the study medication for efficacy analysis after ICEs



## 6.4 SUBJECT SETS ANALYSED

The following patient analysis sets are defined:

• Screened Set (SS): includes all patients who signed informed consent and were screened for the trial with at least one screening procedure done at Visits 1 or 1a.

- Randomised Set (RS): includes all patients who signed informed consent and were randomised into the trial, regardless of whether a patient was treated with trial medication. Patients randomized in error and discontinued from the study before the start of trial medication will be excluded from the RS. Patients in RS will be analysed under the randomized trial medication. The RS will be used for efficacy analyses as well as demographics and baseline characteristics.
- Treated Set (TS): includes all patients who signed informed consent and were treated with at least one dose of the trial medication. Patients in TS will be analysed under the actual trial medication received at randomisation. The TS will be used for safety analyses.
- PK parameter analysis Set (PKS): includes all treated patients who have at least one evaluable PK plasma concentration measurement.
- Ocular sub-study Set (EYE): includes all treated patients who consented to participate in the ocular sub-study (including late/retrospective consent to the ocular sub-study) and had evaluable ophthalmologic measurements. The Ocular sub-study Set will be used for safety analyses, demographics, baseline characteristics and ophthalmologic endpoint analyses of the ocular sub-study.



#### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

Missing or incomplete AE dates will be imputed according to BI standards (1). Missing data and outliers of PK data will be handled according to ( $\underline{2}$ ).

If not specified otherwise, missing data will not be imputed and will remain missing. Potential outliers will be reported and analysed as observed.

Handling and derivation of total/domain/subscale scores for the assessment scales in case of missing individual item scores are specified below:

#### **MCCB**

Handling of missing data in MCCB tests will follow the MCCB Manual (available in the ISF). See Section 10.1 for detailed descriptions and imputation rules.

#### **SCoRS**

For the 20-item SCoRS assessment, if six or more of the 20 items have missing response, which includes the response of "N/A", for a subject at a visit, then the SCoRS total score for that subject at that visit is missing. If five or less of the 20 items have missing response, which includes the response of "N/A", for a subject at a visit, then the item with missing response will be imputed first with the average of the non-missing item values for the subject at the visit, and then SCoRS total score for the subject at the visit will be derived as the sum of the non-missing item values and the imputed item values.

#### **PANSS**

PANSS total and subscale scores will be calculated as sums of their constituting item scores. If  $\leq 20\%$  of the items are missing in the calculation of the total or subscale scores, the missing items will be temporarily imputed with the mean of the non-missing item scores. The total or subscale score will then be calculated as the sum of the non-missing and imputed item scores.

For calculation of PANSS total score and the subscale scores, the maximum numbers of missing items allowed are:

| PANSS total score: | 6 out of 30 |
|--------------------------------------------------|-------------|
| Positive Symptom: | 1 out of 7 |
| Negative Symptom: | 1 out of 7 |
| General Psychopathology: | 3 out of 16 |
| Marder Positive Factor: | 1 out of 8 |
| Marder Disorganized Thought Factor: | 1 out of 7 |
| Marder Negative Factor: | 1 out of 7 |
| Marder Uncontrolled Hostility/Excitement Factor: | 0 out of 4 |
| Marder Anxiety/Depression Factor: | 0 out of 4 |

If more than the maximum allowed number of items are missing, the score will not be calculated.

#### **PRECIS**

PRECIS total score and domain scores will be calculated as averages of their constituting non-missing items. <u>Table 6.6:1</u> lists the minimum number of non-missing items required for

calculation of PRECIS total score and domain scores. If fewer items than the minimum requirement are non-missing, the corresponding total score or domain score will not be calculated and will be treated as missing.

Table 6.6: 1 PRECIS minimum non-missing items required for total/domain score calculation

| | | Minimum required non-missing items |
|--------------------|--------------------|------------------------------------|
| | | PRECIS (28-item version) |
| | Memory | 3 out of 6 |
| | Communication | 3 out of 4 |
| Domain | Self-Control | 3 out of 3 |
| Don | Executive Function | 4 out of 4 |
| | Attention | 3 out of 6 |
| | Sharp Thinking | 3 out of 3 |
| PRECIS total score | | 19 out of 26 |

#### 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

In general, baseline values are the measurements taken prior to the first administration of trial medication. For assessments of efficacy, PANSS and C-SSRS, baseline will be defined as the last available assessment performed at or before randomization (Visit 2), and no later than the day of the first administration of study medication. Assessments done at Visit 1 or Visit 1a can be used as baseline if Visit 2 assessment is not planned, not available, or invalid.

For MCCB, only the assessment performed at randomization (Visit 2), and no later than the day of the first administration of study medication will be used as the baseline. If no valid assessment is available at Visit 2 then baseline value will be missing; assessments performed at Visits 1 and 1a will not be used as baseline.

Tables in this section define the analysis visits and windows which will be used for the analyses of efficacy and safety endpoints. Actual study day will be calculated starting with the date of first administration of trial treatment as Day 1. Unscheduled assessments will be mapped to the analysis visits together with the scheduled assessments.

Inclusion of an assessment into mapping consideration will depend on its on-/off-treatment status and per specific estimand (i.e., off-treatment data will be included into mapping consideration only when the associated ICE is handled under the treatment policy approach). If more than one assessment falls into the same analysis visit window, the assessment performed closest to the planned day will be selected for analyses. In case of a tie, the later assessment will be used.

Table 6.7: 1 Analysis visit windows for MCCB, VRFCAT, SCoRS, and PANSS

| Analysis Visit | Nominal Week | Planned Day | Actual Day Window |
|----------------|--------------|-------------|-------------------|
| Baseline | | 1 | ≤1 |
| Visit 6 | Week 12 | 85 | 2 – 126 |
| Visit 11 | Week 26 | 183 | ≥127 |

Table 6.7: 2 Analysis visit windows for PRECIS, EQ-5D-5L (patient)

| Analysis Visit | Nominal Week | Planned Day | Actual Day Window |
|----------------|--------------|-------------|-------------------|
| Baseline | | 1 | ≤1 |
| Visit 7 | Week 15 | 106 | 2 – 126 |
| Visit 10 | Week 24 | 169 | ≥127 |

Table 6.7: 3 Analysis visit windows for Tower of London, SDS, EQ-5D-5L (caregiver), SPGI-S, SCQ

| Analysis Visit | Nominal Week | Planned Day | Actual Day Window |
|---|---|---|---|
| Baseline | | 1 | ≤1 |
| Visit 10 (for SDS only) | Week 24 | 169 | ≥2 |
| Visit 11<br>(for Tower of London, EQ-5D-<br>5L (caregiver), SPGI-S, and<br>SCQ) | Week 26 | 183 | ≥2 |

Table 6.7: 4 Analysis visit windows for CGI-S

| Analysis Visit | Nominal Week | Planned Day | Actual Day Window |
|----------------|--------------|-------------|-------------------|
| Baseline | | 1 | ≤1 |
| Visit 6 | Week 12 | 85 | 2 – 126 |
| Visit 10 | Week 24 | 169 | 127 – 175 |
| Visit 11 | Week 26 | 183 | ≥176 |

Table 6.7: 5 Analysis visit windows for PGI-S

| Analysis Visit | Nominal Week | Planned Day | Actual Day Window |
|----------------|--------------|-------------|-------------------|
| Baseline | | 1 | ≤1 |
| Visit 10 | Week 24 | 169 | 2 – 175 |
| Visit 11 | Week 26 | 183 | ≥176 |

Table 6.7: 6 Analysis visit windows for SAS/BARS/AIMS

| Analysis Visit | Nominal Week | Planned Day | Actual Day Window |
|----------------|--------------|-------------|-------------------|
| Baseline | | 1 | ≤1 |
| Visit 4 | Week 6 | 43 | 2 – 74 |
| Visit 7 | Week 15 | 106 | 75 – 137 |
| Visit 10 | Week 24 | 169 | 138 – 175 |
| Visit 11 | Week 26 | 183 | ≥176 |

Table 6.7: 7 Analysis visit windows for clinical laboratory evaluations (on-treatment period)

| Analysis Visit | Nominal Week | Planned Day | Actual Day Window |
|----------------|------------------------|-------------|-------------------|
| Baseline | | 1 | ≤1 |
| Visit 2 | Week 0 (post-baseline) | 1 | 2 – 35 |
| Visit 4 | Week 6 | 43 | 36 – 77 |
| Visit 6 | Week 12 | 85 | 78 – 119 |
| Visit 8 | Week 18 | 127 | 120 – 140 |
| Visit 9 | Week 21 | 148 | 141 – 161 |
| Visit 10 | Week 24 | 169 | 162 – 175 |
| Visit 11 | Week 26 | 183 | ≥176 |

All post-baseline actual day windows will be curtained at the end of residual period if earlier than the specified upper bound in the table.

Table 6.7: 8 Analysis visit windows for weight and vital signs (on-treatment period)

| Analysis Visit | Nominal Week | Planned Day | Actual Day Window |
|----------------|------------------------|-------------|-------------------|
| Baseline | | 1 | ≤1 |
| Visit 2 | Week 0 (post-baseline) | 1 | 2 – 56 |
| Visit 5 | Week 9 | 64 | 57 – 119 |
| Visit 8 | Week 18 | 127 | 120–175 |
| Visit 11 | Week 26 | 183 | ≥176 |

All post-baseline actual day windows will be curtained at the end of residual period if earlier than the specified upper bound in the table.

Table 6.7: 9 Analysis visit windows for Ophthalmological variables

| Analysis Visit | Nominal Week | Planned Day | Actual Day Window |
|----------------|--------------|-------------|-------------------|
| Baseline | | -7 | ≤1 |
| Visit 10 | Week 24 | 169 | ≥2 |

Note that for placebo patients who rolled over to the extension study, any ophthalmological assessments incidentally performed after the first administration of iclepertin in the extension study will not be included in the safety analysis.

#### 7. PLANNED ANALYSIS

For End-Of-Text tables, the set of summary statistics is: N / Mean / Standard Deviation (STD) / Min / Median / Max.

For tables that are provided for endpoints with some extreme data, median, quartiles and percentiles are preferred to mean, standard deviation, minimum and maximum.

In general, means, medians, and percentiles are presented to one more decimal place than the raw data and STDs are presented to two more decimal places than the raw data. Minima and Maxima are presented to the same number of decimal places as the raw data.

Tabulations of frequencies for categorical data include all possible categories (even if there is no count in a category) and display the number of observations in a category as well as the percentage (%) relative to the number of subjects in the respective treatment group (unless otherwise specified, all subjects in the respective subject set whether they have non-missing values or not). Percentages are rounded to one decimal place, unless the denominator is smaller than 100 (in all treatment columns), in which case percentages are rounded to the nearest integer. The category missing will be displayed only if there are actually missing values.

If a table presents only categorical data, "[N (%)]" is displayed in the column header only.

Abbreviations (e.g. Wors.) or acronyms (e.g. PD) will not be displayed in tables and subject data listings without any explanation. They will be either spelled out or explained in footnotes.

If applicable, days will be converted to weeks, months or years as follows:

- weeks = days  $\div$  7
- months =  $12 \times \text{days} \div 365.25$
- years = days  $\div$  365.25

#### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the report.

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

Only descriptive statistics are planned for this section of the report.

Concomitant diseases will be coded similarly as AEs based on the most current MedDRA version. A summary of concomitant diseases will be provided by treatment group, system organ class (SOC), and preferred term (PT).

Concomitant therapies (CTs) will be coded according to WHO DD and classified by the Anatomical, Therapeutic, Chemical (ATC) classification system. The third ATC level will be

used to categorise CTs by therapy type. In situations where a medical product may be used for more than one equally important indication, there are often several classification alternatives. As appropriate, subjects receiving CTs with more than one possible ATC level-three category will be counted more than once. CTs will be summarised in two groups: CNS-active and non-CNS-active concomitant medications.

Summaries will also be provided for the following CTs of special interest: antipsychotics, benzodiazepines, anticholinergics, antiepileptics, and antidepressants, as defined in <u>Table 10.7: 1</u>.

#### 7.3 TREATMENT COMPLIANCE

Only descriptive statistics are planned for this section of the report. See <u>Section 5.4</u> for definitions of treatment compliance. In addition, descriptive statistics of treatment adherence based on the AiCure data, as defined in <u>Section 5.4</u>, will also be reported.

#### 7.4 PRIMARY ENDPOINT ANALYSIS

#### 7.4.1 Primary analysis

In the primary analysis under the primary estimand, intercurrent events will be addressed using a strategy that differs depending upon the nature of the intercurrent event. For details please refer to Section 6.3 above (or Section 7 of the CTP). This primary analysis of the primary efficacy endpoint will be performed on the Randomized Set. With regard to the stratification factor, subjects will be analyzed according to the screening MCCB overall composite T-score stratum to which they correctly belong. Missing data resulting from the strategy (including both actual missing outcomes and excluded outcomes) will be handled using a mixed-effects model for repeated measures (MMRM) under the assumption of missing at random.

The primary endpoint is the change from baseline to Week 26 in overall composite T-score of the MCCB.

The primary analysis will be a restricted maximum likelihood (REML) based approach using a mixed-effects model for repeated measurements (MMRM) comparing the change from baseline in MCCB overall composite T-score at Week 26 between iclepertin 10 mg QD and placebo. The MMRM will includes the fixed categorical effects of treatment at each visit, a fixed categorical effect of the stratification factor using the screening MCCB overall composite T-score, and a fixed effect for the continuous covariate of baseline (i.e. baseline MCCB overall composite T-score) at each visit. Visit will be treated as the repeated measure with an unstructured covariance structure used to model the within-subject dependencies.

The statistical model will be as follows:

$$y_{ijkm} = \beta_j S_i + \tau_{jk} + \varphi_m + e_{ij},$$

where

$$(e_{i1}, \ldots, e_{iJ})' \sim N_J(\mathbf{0}, \Sigma),$$

and

```
y_{ijkm}= response variable for subject i in stratum m at visit j randomized to treatment k S_i= the baseline MCCB overall composite T-score of subject i,i=1,2,... \beta_j= coefficient of baseline effect at visit j,j=1,...,J \tau_{jk}= the effect of treatment k at vist j,k=1,2 \varphi_m= the effect of screening MCCB overall composite T-score stratum m for m=1,2, and \varphi_1\equiv 0 for stratum 1 of T-score <30 e_{ij}= the random error associated with jth visit of the ith subject. \Sigma= a J\times J unstructured covariance matrix
```

The Kenward-Roger approximation will be used to estimate the denominator degrees of freedom and adjust standard errors. Significance tests will be based on least-squares means, following the testing strategy described in CTP Section 7.1. The primary treatment comparison will be the contrast between iclepertin 10 mg QD and placebo at Week 26. Results of the MMRM (N, mean, SE and 95% CI per dose group and timepoint) will be presented in tables and displayed graphically.

Example SAS code for the primary analysis of MMRM is provided in <u>Section 10.2.1</u>. In the event of non-convergence, methods described in <u>Section 10.2.2</u> will be attempted to overcome the issue.







#### 7.5 SECONDARY ENDPOINT ANALYSIS

## 7.5.1 Key secondary endpoint analysis

## 7.5.1.1 Primary analysis

For the two key secondary efficacy endpoints of change from baseline at Week 26 in SCoRS interviewer total score and VRFCAT adjusted total time T-score, the same strategy for handling the intercurrent events in the primary analysis under the primary estimand will be applied.

The primary analysis will be a restricted maximum likelihood (REML) based approach using the same primary analysis model of MMRM specified in <u>Section 7.4.1</u>, but with the baseline covariate replaced by the baseline of the corresponding key secondary endpoint.





## 7.5.2 (Other) Secondary endpoint analysis

For the secondary efficacy endpoints of change from screening to Week 24 in PRECIS total score and change from baseline to Week 26 in Tower of London number of correct responses T-score, the same strategy for handling the intercurrent events in the primary analysis under the primary estimand will be applied.

For change from screening to Week 24 in PRECIS total score, the primary analysis will be a restricted maximum likelihood (REML) based approach using the same primary analysis model of MMRM specified in Section 7.4.1, but with the baseline covariate replaced by the screening PRECIS total score. The same subgroup analyses as planned for the primary efficacy endpoint in Section 7.4.3 will also be conducted for PRECIS total score.

For change from baseline to Week 26 in the T-score of number of correct responses on Tower of London, an analysis of covariance (ANCOVA) model including treatment, stratification factor of screening MCCB overall composite T-score (<30, ≥30), and baseline number of correct responses on Tower of London T-score will be fitted to the data.





#### 7.7 EXTENT OF EXPOSURE

Extent of exposure will be summarized for the treated set using descriptive statistics for days on treatment as well as frequency and percentage of subjects in the following categories: <42, 42 - <84, 84 - <126, 126 - <168, 168 - <179, 179 - <190,  $\ge 190$ .

#### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the treated set and other subject sets as appropriate.

#### 7.8.1 Adverse events

Unless otherwise specified, the analyses of AEs will be descriptive in nature. All analyses of AEs will be based on the number of subjects with AEs and not on the number of AEs. The reporting and analyses of AEs will follow the BI guideline (3). AEs will be coded with the most current version of MedDRA®.

For further details on summarization of AE data, please refer to (1, 3).

The analysis of AEs will be based on the concept of treatment emergent AEs. That means that all AEs occurring between the date of the first administration of trial treatment till the date of the last administration of trial treatment + residual effect period will be assigned to the ontreatment period. All AEs occurring before the first administration of trial treatment will be assigned to 'screening' and all AEs occurring after the residual effect period will be assigned to 'follow-up'. For details on the treatment definition, see Section 6.1.

## Adverse events of special interest (AESIs)

A hepatic injury is defined by the following alterations of hepatic laboratory parameters:

- an elevation of AST and / or ALT  $\geq$  3 fold ULN combined with an elevation of total bilirubin  $\geq$  2 fold ULN measured in the same blood draw sample; and / or
- marked peak aminotransferase (ALT and / or AST) elevations  $\geq 10$  fold ULN.

See CTP Section 5.2.6.1.

# Other significant AEs

| <b>User-defined AE category</b> | MedDRA preferred terms | |
|---|---|---|
| Drug abuse, dependence, | Accidental death | Intentional overdose |
| withdrawal and substance-<br>related disorders, including | Drug abuse | Muscle rigidity |
| diversion | Accidental overdose | Nasal necrosis |
| | Accidental poisoning | Nasal septum perforation |
| | Dependence | Nasal septum ulceration |
| | Drug abuser | Needle track marks |
| | Product administered at | Neonatal complications of substance |
| | inappropriate site | abuse |
| | Drug dependence | Overdose |
| | Drug detoxification | Poisoning |
| | Drug dependence antepartum | Poisoning deliberate |
| | Drug dependence, postpartum | Substance dependence |
| | Drug diversion | Prescription form tampering |
| | Drug tolerance | Product tampering |
| | Drug tolerance increased | Product used for unknown indication |
| | Toxicity to various agents | Rebound effect |
| | Drug use disorder | Seizure |
| | Drug use disorder antepartum | Status epilepticus |
| | Drug use disorder, postpartum | Substance abuse |
| | Drug withdrawal convulsions | Substance abuser |
| | Drug withdrawal headache | Substance use |
| | Drug withdrawal syndrome | Substance use disorder |
| | Drug withdrawal syndrome neonatal | Substance-induced mood disorder |
| | Generalised tonic-clonic seizure | Substance-induced psychotic disorder |
| | Hangover | Treatment noncompliance |
| | Intentional product misuse | Withdrawal syndrome |
| Euphoria-related adverse | Dizziness | Feeling drunk |
| events | Euphoric mood | Feeling of relaxation |
| | Feeling abnormal | Inappropriate affect |
| CNS depressant effects | Depressed level of consciousness | Sedation |
| | Fatigue | Sluggishness |
| | Hypersomnia | Somnolence |
| | Lethargy | Stupor |
| | Loss of consciousness | |
| Stimulation and anxiety- | Agitation | Morbid thoughts |
| related adverse events | Anxiety | Nervousness |
| | Anxiety disorder | Panic attack |
| | Anticipatory anxiety | Panic disorder |
| | Energy increased | Panic reaction |
| | Fear | Psychogenic tremor |

| | Fear of death | Psychomotor hyperactivity |
|---|---|---|
| | Feeling jittery | Restlessness |
| | Generalised anxiety disorder | Tension |
| | Hypervigilance | |
| Perceptual disturbances / | Abnormal dreams | Hypoaesthesia |
| psychotomimetic effects | Acute psychosis | Ideas of reference |
| | Aggression | Illogical thinking |
| | Alice in wonderland syndrome | Illusion |
| | Altered state of consciousness | Incoherent |
| | Altered visual depth perception | Indifference |
| | Anger | Jamais vu |
| | Communication disorder | Loose associations |
| | Confusional state | Magical thinking |
| | Consciousness fluctuating | Nightmare |
| | Déjà vu | Paranoia |
| | Delirium | Paroxysmal perceptual alteration |
| | Delusion | Psychotic behaviour |
| | Delusion of grandeur | Psychotic disorder |
| | Delusion of reference | Psychotic symptom |
| | Delusion of replacement | Reactive psychosis |
| | Delusional perception | Rebound psychosis |
| | Derailment | Sensory disturbance |
| | Disinhibition | Sensory level abnormal |
| | Disorientation | Slow speech |
| | Dysarthria | Somatic delusion |
| | Flight of ideas | Somatic hallucination |
| | Formication | Staring |
| | Hallucination | Suspiciousness |
| | Hallucination, auditory | Tangentiality |
| | Hallucination, gustatory | Thinking abnormal |
| | Hallucination, olfactory | Thought blocking |
| | Hallucination, synaesthetic | Thought broadcasting |
| | Hallucination, tactile | Thought insertion |
| | Hallucination, visual | Thought withdrawal |
| | Hallucinations, mixed | Transient psychosis |
| | Hostility | |
| Dissociation | Daydreaming | Hypogeusia |
| | Depersonalisation/derealisation disorder | Metamorphopsia |
| | Derealisation | Ocular discomfort |
| | Diplopia | Oral dysaesthesia |
| | Dissociation | Oral hyperaesthesia |

| | Dissociative disorder | Pain threshold decreased |
|---|---|---|
| | Dissociative identity disorder | Paraesthesia |
| | Dysaesthesia | Paraesthesia oral |
| | Dysaesthesia pharynx | Pharyngeal hypoaesthesia |
| | Dysgeusia Dysgeusia | Pharyngeal paraesthesia |
| | Dysmetropsia | Photophobia |
| | Feeling cold | Photopsia |
| | | • |
| | Feeling hot | Synaesthesia |
| | Feeling of body temperature change Flashback | Time perception altered Tinnitus |
| | Hyperacusis | Vision blurred |
| | Hyperaesthesia | Visual impairment |
| | Hypersensitivity | |
| Mood disorders and disturbances | Abnormal behaviour | Depressive delusion |
| | Affect lability | Depressive symptom |
| | Affective disorder | Disturbance in social behaviour |
| | Anhedonia | Emotional disorder |
| | Antisocial behaviour | Emotional distress |
| | Apathy | Feeling of despair |
| | Asocial behaviour | Flat affect |
| | Attention-seeking behaviour | Hypomania |
| | Belligerence | Impatience |
| | Blunted affect | Impulse-control disorder |
| | Compulsive cheek biting | Impulsive behaviour |
| | Compulsive handwashing | Irritability |
| | Compulsive hoarding | Mania |
| | Compulsive lip biting | Mood altered |
| | Compulsive sexual behaviour | Mood swings |
| | Compulsive shopping | Parasomnia |
| | Obsessive-compulsive symptom | Personality change |
| | Compulsions | Sleep talking |
| | Confusional arousal | Sleep terror |
| | Depressed mood | Sleep-related eating disorder |
| | Depression | Somnambulism |
| Mental and cognitive | Amnesia | Impaired driving ability |
| impairment | Amnestic disorder | Impaired reasoning |
| | Anterograde amnesia | Judgement impaired |
| | Balance disorder | Memory impairment |
| | Bradyphrenia | Mental disability |
| | Change in sustained attention | Mental disorder |
| | Cognitive disorder | Mental impairment |
| | Confabulation | Mental status changes |
| | Commonation | 1.1011tai batab cilaligos |
| Coordination abnormal | Paramnesia |
|--------------------------|-----------------------------|
| Distractibility | Psychomotor retardation |
| Disturbance in attention | Psychomotor skills impaired |
| Dyslogia | Retrograde amnesia |
| Executive dysfunction | Transient global amnesia |

According to ICH E3, in addition to deaths and serious adverse events, 'other significant' AEs need to be listed in the clinical trial report. These will include:

- 1. Any adverse events that led to an intervention, such as withdrawal of drug treatment.
- 2. Marked haematological and other lab abnormalities or lead to significant concomitant therapy as identified by the Clinical Monitor/Investigator during medical quality review at TOM.

#### AEs suggestive of abuse potential or related to CNS depressant effects

In support of an evaluation of human abuse potential, user-defined AE categories (UDAEC) are defined in <u>Table 7.8.1: 1</u> for AEs suggestive of abuse potential and AEs related to CNS depressant effects.

Table 7.8.1: 1 MedDRA preferred terms for user-defined AE categories of AEs suggestive of abuse potential or related to CNS depressant effects

Other UDAECs are defined as follow:

#### Ocular events

The grouping of "ocular events" includes all MedDRA preferred terms under the SOC of "eye disorder" regardless of primary or secondary SOC.

#### Anaemia

Anaemia will be analyzed by BI customized medical query (BIcMQ) of Decreased haemoglobin and anaemia (incl. non-haematological causes), as defined in Table 7.8.1: 2

In addition, Standardised MedDRA Query (SMQ) of Haematopoietic cytopenias will be analyzed.

Table 7.8.1: 2 MedDRA preferred terms for BIcMQ of Decreased haemoglobin and anaemia (incl. non-haematological causes)

| User-defined AE category | MedDRA preferred terms | |
|---|---|---|
| Decreased haemoglobin and anaemia (incl. non-haematological causes) | Anaemia | Haemoglobin abnormal |
| | Anaemia Heinz body | Haemoglobin decreased |
| | Anaemia folate deficiency | Haemolytic anaemia |
| | Anaemia macrocytic | Haemolytic anaemia enzyme specific |
| | Anaemia megaloblastic | Haemolytic icteroanaemia |
| | Anaemia of chronic disease | Hyperchromic anaemia |
| | Anaemia of malignant disease | Hypochromic anaemia |

| Anaemia postoperative | Hypoplastic anaemia |
|------------------------------------|-------------------------------------|
| Anaemia splenic | Iron deficiency anaemia |
| Anaemia vitamin B12 deficiency | Leukoerythroblastic anaemia |
| Anaemia vitamin B6 deficiency | Macrocytosis |
| Anaemic hypoxia | Melanaemia |
| Anaemic retinopathy | Microangiopathic haemolytic anaemia |
| Aplasia pure red cell | Microcytic anaemia |
| Aplastic anaemia | Nephrogenic anaemia |
| Autoimmune anaemia | Normochromic anaemia |
| Autoimmune aplastic anaemia | Normochromic normocytic anaemia |
| Autoimmune haemolytic anaemia | Normocytic anaemia |
| Blood loss anaemia | Pernicious anaemia |
| Cardiac haemolytic anaemia | Proerythroblast count abnormal |
| Cold type haemolytic anaemia | Proerythroblast count decreased |
| Coombs negative haemolytic anaemia | Protein deficiency anaemia |
| Coombs positive haemolytic anaemia | Radiation anaemia |
| Copper deficiency anaemia | Red blood cell abnormality |
| Deficiency anaemia | Red blood cell count abnormal |
| Dilutional anaemia | Red blood cell count decreased |
| Erythroblast count abnormal | Reticulocyte count abnormal |
| Erythroblast count decreased | Reticulocyte count decreased |
| Erythroid dysplasia | Reticulocyte percentage decreased |
| Erythroid maturation arrest | Reticulocytopenia |
| Erythropenia | Scorbutic anaemia |
| Erythropoiesis abnormal | Sideroblastic anaemia |
| Erythropoietin deficiency anaemia | Spherocytic anaemia |
| Haematocrit abnormal | Spur cell anaemia |
| Haematocrit decreased | Warm autoimmune haemolytic anaemia |

# **Drowsiness**

Drowsiness will be analyzed by a customized query defined in <u>Table 7.8.1: 3</u>.

Table 7.8.1: 3 MedDRA preferred terms for user-defined AE category of Drowsiness

| User-defined AE category | MedDRA preferred terms | Scope |
|--------------------------|----------------------------------|--------|
| Drowsiness | Depressed level of consciousness | Narrow |

| Post-injection delirium sedation syndrome | Narrow |
|-------------------------------------------|--------|
| Radiation somnolence syndrome | Narrow |
| Sedation | Narrow |
| Altered state of consciousness | Broad |
| Brain fog | Broad |
| Concussion | Broad |
| Consciousness fluctuating | Broad |
| Intracranial hypotension | Broad |
| Lethargy | Broad |
| Obstructive sleep apnoea syndrome | Broad |
| Orexin deficiency | Broad |
| Pickwickian syndrome | Broad |
| Post concussion syndrome | Broad |
| Presyncope | Broad |
| Sedation complication | Broad |
| Sleep-related hypoventilation | Broad |
| Shift work disorder | Broad |
| Sleep apnoea syndrome | Broad |

## Sleep disorder

Sleep disorder related AE search terms are based upon the FDA Medical Queries (FMQs) of Insomnia (broad) and Somnolence (broad). Refer to <u>Table 7.8.1: 4</u> for a list of MedDRA preferred terms in each of the groupings.

Table 7.8.1: 4 MedDRA preferred terms for user-defined AE categories of sleep disorder AEs

| User-defined AE category | MedDRA preferred terms | |
|---|---|---|
| FMQ Insomnia (broad) | Advanced sleep phase | Primary insomnia |
| | Behavioural induced insufficient sleep syndrome | Psychophysiologic insomnia |
| | Circadian rhythm sleep disorder | Shift work disorder |
| | Delayed sleep phase | Sleep disorder due to general medical condition, insomnia type |
| | Dyssomnia | Sleep disorder due to general medical condition, mixed type |
| | Early morning awakening | Terminal insomnia |
| | Fatal familial insomnia | Dysfunctions associated with sleep stages or arousal from sleep |
| | Hyposomnia | Dyssomnia NOS |
| | Initial insomnia | Jet lag |
| | Insomnia | Microsleep |
| | Insomnia exacerbated | Sleep deficit |
| | Insomnia NEC | Sleep disorder |
| | Insomnia related to another mental condition | Sleep disorder due to a general medical condition |
| | Irregular sleep phase | Sleep disorder NOS |
| | Irregular sleep wake rhythm disorder | Sleep disorder therapy |

| | Middle insomnia | Sleep inertia |
|---|---|---|
| | Non-24-hour sleep-wake disorder | Sleep study abnormal |
| | Poor quality sleep | |
| FMQ Somnolence (broad) | Central nervous system depression NOS | Sedation aggravated |
| | Consciousness fluctuating | Somnolence |
| | Depressed level of consciousness | Somnolence neonatal |
| | Hypersomnia | Stupor |
| | Infant sedation | Altered state of consciousness |
| | Lethargy | Fatigue |
| | Neonatal oversedation | Fatigue aggravated |
| | Primary hypersomnia | Prostration |
| | Sedation | Sluggishness |

An overall summary of adverse events will be presented, including frequency of schizophrenia relapse. The frequency of subjects with AEs will be summarised by treatment, primary system organ class (SOC) and preferred term (PT). The SOCs will be sorted by default in descending frequency and PTs will be sorted in descending frequency within an SOC in the iclepertin arm. Separate tables will be provided for patients with

- Related AEs
- Serious AEs
- Serious related AEs
- AESIs
- Other significant AEs
- AEs leading to death
- AE leading to discontinuation of trial medication
- AEs occurred with incidence in the preferred term >2%
- AEs suggestive of abuse potential or related to CNS depressant effects
- AEs in user-defined AE categories
- AEs occurred during the follow-up period.

## 7.8.2 Laboratory data

The analyses of laboratory data will be descriptive in nature and will follow BI standards (4).

Descriptive statistics for laboratory values will be displayed using the converted values in standard unit for data analyzed by the central laboratory. Shift tables of change in laboratory measurements between baseline and minimum, maximum or last value on treatment will be presented.

#### 7.8.3 Vital signs

Only descriptive statistics are planned for this section of the report.

#### 7.8.4 ECG

Clinically relevant abnormal ECG findings will be reported and analysed as AEs.

#### 7.9 OTHER ANALYSES

Population pharmacokinetic and pharmacokinetic/pharmacodynamic analyses

A population PK analysis for iclepertin may be performed. Data of this study may be pooled with data of other iclepertin trials. Population PK and PK/PD analyses will be subject to a separate analysis plan(s) and report(s), and will not be part of the CTR.

### Ophthalmologic variables

Each ophthalmologic variable is measured for both the right eye and the left eye. For continuous variables, summary statistics including mean, median, standard deviation, minimum, maximum will be presented for the change from baseline measurements.

For categorical variables, shift tables will be presented for the categorical changes from baseline.

# 8. TIMEPOINT OF RELEASE OF TREATMENT INFORMATION

The treatment information will be released to unblind the trial database after the last patient has completed their End-of-Study/Follow-up visit and all data has been entered and cleaned as defined in the "Data Ready to be Unblinded and/or Final Trial Closure Notification" (RUN) form.

# 9. REFERENCES

| 1. | BI-KMED-BDS-HTG-0035: "How to Guide: Handling of Missing and Incomplete AE dates", current version, KMED |
|---|---|
| 2. | <i>BI-KMED-TMCP-HTG-0025:</i> "How to Guide: Standards and Processes for Analyses Performed within Clinical Pharmacokinetics/Pharmacodynamics", current version, KMED. |
| 3. | BI-KMED-BDS-HTG-0041: "How to Guide: Analysis and Presentation of AE Data from Clinical Trials", current version, KMED |
| 4. | BI-KMED-BDS-HTG-0042: "How to Guide: Handling, Display and Analysis of Laboratory Data", current version, KMED |
| 5. | Keefe et al. (2017) Placebo Response and Practice Effects in Schizophrenia Cognition Trial. JAMA Psychiatry 74(8):807-814. [R19-3822] |
| 6. | Carpenter, J. and Kenward, M. (2013) Multiple Imputation and its Application, 1st ed. Wiley, New York. [R22-0188] |
| 7. | Liu, F. and Peng, L. (2016) On analysis of longitudinal clinical trials with missing data using reference-based imputation. Journal of Biopharmaceutical Statistics, 26(5):924-936. [R23-1692] |
| 8. | Guizzaro, et al (2021) The Use of a Variable Representing Compliance Improves Accuracy of Estimation of the Effect of Treatment Allocation Regardless of Discontinuation in Trials with Incomplete Follow-up. Statistics in Biopharmaceutical Research, 13(1):119-127. [R23-1510] |
| 9. | Little, R. J. & Rubin, D. B. (2002). Statistical Analysis with Missing Data (2nd ed). New York: John Wiley & Sons. [R12-2094] |
| 10. | Bell, J. (2022). Implementation of the treatment policy strategy for continuous longitudinal endpoints: a comparison of estimation methods. PSI Conf, Gothenburg. [R23-0137] |















## Boehringer Ingelheim TSAP for BI Trial No: 1346.11

 c44703258-02

#### **HISTORY TABLE** 11.

Table 11: 1 History table

| Version | Date<br>(DD-MMM-<br>YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|
| 2 | 25-OCT-24 | | Table 7.8.1: 2 | This table was updated to fix a truncation issue in the previous version. |